CLINICAL TRIAL: NCT05442385
Title: Patterns and Outcome of Cardiac Patients Admitted to PICU
Brief Title: Indication of Admission , Treatment and Outcomes of Cardiac Patients in PICU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Refaet Zakher, principal investigator, Assiut University
Other Study IDs: cardiac patient in PICU
Record Dates: First submitted 2022-06-17; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiac patients admitted to PICU: To describe the clinical patterns of infants and children with cardiac disease admitted to PICU and their outcome.
  Interventions: Other: Evidence based management

INTERVENTIONS:
Other: Evidence based management — clinical patterns , laboratory investigations , radiology , lines of managements and outcome of each modality of treatment

SUMMARY:
Aim of the work:

To describe the clinical patterns criteria of infants and children with cardiac disease admitted to PICU and their outcome.

DETAILED DESCRIPTION:
Intensive care has become very important in the management of critically ill children. The pediatric intensive care unit (PICU) is a part of the hospital where critically ill pediatric patients who require advanced airway, respiratory, and hemodynamic supports are usually admitted with the aim of achieving an outcome better than if the patients were admitted into other parts of the hospital. The care of critically ill children remains one of the most demanding and challenging aspects of the field of pediatrics. The main purpose of the PICU is to prevent mortality by intensively monitoring and treating critically ill children who are considered at high risk of mortality. This, however, comes at a huge cost to all the parties involved the hospital, the personnel, and the care givers of patients. It is usually only offered to patients whose condition is potentially reversible and who have a good chance of surviving with intensive care support. Since these patients are critically ill, the outcome of intervention is sometimes difficult to predict. In critical care medicine, intensive care unit (ICU) results can be assessed on the basis of outcomes such as "death" or "survival" by means of indicators such as mortality rates. Evaluation of the outcomes of medical interventions can assess the efficacy of treatment, making it possible to take better decisions, to further improve quality of care, to standardize conduct, and to ensure effective management of the high-level resources needed to deliver intensive care services thereby optimizing resource utilization. Although mortality in patients depends on many factors such as demographic and clinical characteristic of population, infrastructure and non-medical factors (management and organization), case mix, and admission practice, it is also affected by ICU performance.

The PICU concept was initially developed about 40 years ago with the first consensus conference on critical care admission held in 1983 by the National Institute of Health in the US The principle that emerged from this group continues to be relevant even today as it identifies patients who should be admitted to the PICU as those who "reversible medical conditions with a reasonable prospect of substantial recovery" Clinical diagnosis model based PICU admission criteria Cardiac conditions cardiogenic shock, myocardial dysfunction: infectious and other complex dysrhythmias requiring close monitoring and intervention, including new onset complete heart block and after cardioversion, acute congestive heart failure requiring hemodynamic support, hypertensive emergencies after cardiac arrest and post-resuscitation, aortic dissection congenital heart disease with cardiopulmonary instability patients presenting to the emergency department with cardiorespiratory or neurologic compromise after high risk intrathoracic or cardiac procedures, need for invasive cardiac monitoring, need for cardiac pacing, pericardial effusion requiring drainage, signs of tamponade ,hypertensive urgency.

Thus it is very important to have clear time sensitive goals in ICU management of these fragile infants and children to minimize mortality and neuromorbidity

ELIGIBILITY:
Inclusion Criteria:

1. Infants and children aged 1 month to 18 years.
2. Patients with primary cardiac diseases either congenital heart disease such VSD or acquired heart disease like rheumatic heart disease and heart failure Admitted to ICU

Exclusion Criteria:

pediatric patient without cardiac diseases

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric cardiac patients aged 1 minth to 18 years old admitted to PICU
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
outcome of Cardiac patients admitted to PICU | Baseline
  To describe the indication of admission and treatment given such as use of inotropes such as epinephrine norepinephrine and mechanical ventilation , high flow nasal canula ..etc and outcome of each case measured by using vital signs (heart rate , Respiratory rate , temperature and blood pressure ) conscious level , signs of heart failure and finally number of deaths

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Lotfy Mohamad Ibrahim, Ass. prof, Study Director — Pediatrics

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bone RC, McElwee NE, Eubanks DH, Gluck EH. Analysis of indications for intensive care unit admission. Clinical efficacy assessment project: American College of Physicians. Chest. 1993 Dec;104(6):1806-11. doi: 10.1378/chest.104.6.1806. PMID 8252969
- [Background] Critical care medicine. JAMA. 1983 Aug 12;250(6):798-804. No abstract available. PMID 6348315
- [Background] Kollef MH, Schuster DP. Predicting intensive care unit outcome with scoring systems. Underlying concepts and principles. Crit Care Clin. 1994 Jan;10(1):1-18. PMID 8118722
- [Background] Nates JL, Nunnally M, Kleinpell R, Blosser S, Goldner J, Birriel B, Fowler CS, Byrum D, Miles WS, Bailey H, Sprung CL. ICU Admission, Discharge, and Triage Guidelines: A Framework to Enhance Clinical Operations, Development of Institutional Policies, and Further Research. Crit Care Med. 2016 Aug;44(8):1553-602. doi: 10.1097/CCM.0000000000001856. PMID 27428118
- [Background] Smith G, Nielsen M. ABC of intensive care. Criteria for admission. BMJ. 1999 Jun 5;318(7197):1544-7. doi: 10.1136/bmj.318.7197.1544. No abstract available. PMID 10356016
- [Background] Carcillo JA, Kuch BA, Han YY, Day S, Greenwald BM, McCloskey KA, Pearson-Shaver AL, Orr RA. Mortality and functional morbidity after use of PALS/APLS by community physicians. Pediatrics. 2009 Aug;124(2):500-8. doi: 10.1542/peds.2008-1967. Epub 2009 Jul 27. PMID 19651576
- [Background] Levin DL, Downes JJ, Todres ID. History of pediatric critical care medicine. J Pediatr Intensive Care. 2013 Dec;2(4):147-167. doi: 10.3233/PIC-13068. PMID 31214438
- [Background] Fiser DH. Outcome evaluations as measures of quality in pediatric intensive care. Pediatr Clin North Am. 1994 Dec;41(6):1423-38. doi: 10.1016/s0031-3955(16)38880-0. PMID 7984393
- [Background] Bertolini G, Ripamonti D, Cattaneo A, Apolone G. Pediatric risk of mortality: an assessment of its performance in a sample of 26 Italian intensive care units. Crit Care Med. 1998 Aug;26(8):1427-32. doi: 10.1097/00003246-199808000-00031. PMID 9710104
- [Background] Lalitha AV, Fassl B, Gist RE, Shah BR, Chawla N, Singh A, Baranawal A, Shamarao S, Vanaki R, Mahajan P, Patel R, Chauhan V, Batra P, Saha A, Galwankar S, Soans S. 2019 WACEM - Academic College of Emergency Experts Consensus Recommendations on Admission Criteria to Pediatric Intensive Care Unit from the Emergency Departments in India. J Emerg Trauma Shock. 2019 Apr-Jun;12(2):155-162. doi: 10.4103/JETS.JETS_140_18. PMID 31198285
- [Background] Frankel LR, Hsu BS, Yeh TS, Simone S, Agus MSD, Arca MJ, Coss-Bu JA, Fallat ME, Foland J, Gadepalli S, Gayle MO, Harmon LA, Hill V, Joseph CA, Kessel AD, Kissoon N, Moss M, Mysore MR, Papo ME, Rajzer-Wakeham KL, Rice TB, Rosenberg DL, Wakeham MK, Conway EE Jr; Voting Panel. Criteria for Critical Care Infants and Children: PICU Admission, Discharge, and Triage Practice Statement and Levels of Care Guidance. Pediatr Crit Care Med. 2019 Sep;20(9):847-887. doi: 10.1097/PCC.0000000000001963. PMID 31483379